CLINICAL TRIAL: NCT01188369
Title: Effects of Levosimendan on Systolic Deformation and Diastolic Function in Patients Eligible for Aortic Valve Replacement With Left Ventricular Hypertrophy
Brief Title: Effects of Levosimendan in Patients Eligible for Aortic Valve Replacement With Left Ventricular Hypertrophy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated prematurely due to high incidence of postoperative atrial fibrillation.
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1616
Record Dates: First submitted 2010-08-10; First posted 2010-08-25 (Estimated); Results first posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2012-08

CONDITIONS: Diastolic Dysfunction; Left Ventricular Hypertrophy
Keywords: levosimendan; heart failure; inotropics; diastolic dysfunction; left ventricular hypertrophy; aortic valve stenosis
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Heart Failure; Aortic Valve Stenosis | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- levosimendan (Experimental): infusion 0,1ug/kg/min for duration of ca. 4 hours prior to operation and until the end of operation
  Interventions: Drug: levosimendan
- Placebo (Placebo Comparator): Identical placebo
  Interventions: Drug: placebo drug

INTERVENTIONS:
Drug: levosimendan — Intravenous infusion, 0,1ug/kg/min, duration 4 hours prior to operation and until the end of operation.
  Other Names: Simdax
  Arms: levosimendan
Drug: placebo drug — Intravenous infusion, colour identical to levosimendan
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a clinical, randomised, double-blinded study in which patients eligible for aortic valve replacement are enrolled. Patients receive infusion of either levosimendan or placebo 4 hours prior to surgery and until the end of surgery.

DETAILED DESCRIPTION:
Levosimendan or placebo will be infusion for approximately 4 hours prior to aortic valve replacement in patients with severe hypertrophy of the left ventricle and echocardiographic signs of diastolic dysfunction. Outcome measures will be obtained at some of the following:

* Approximately 4 hours prior to surgery. Baseline. Start of levosimendan/placebo infusion
* Immediately before surgery
* After induction of anaesthesia and before "knife time" = start of surgery.
* At the end of surgery: Levosimendan infusion will stop.
* Approximately 4 hours after surgery immediately before extubation.
* Approximately 21 hours after surgery
* Approximately 96 hours after surgery (day 4)
* 6 months after surgery

Outcome measures are comprised of invasive measurements, blood samples, transthoracic echocardiography and transoesophageal echocardiography focusing on measures of systolic and diastolic function of the heart.

Interim analysis will be conducted after 30 included patients.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for aortic valve replacement
* EF > 45%
* Left ventricular posterior wall > 12mm
* Sinus rhythm

Exclusion Criteria:

* Concomitant bypass operation
* Severe mitral insufficiency
* Active endocarditis
* Insufficient ultrasound opportunity
* Systolic blood pressure < 100 mmHg
* moderate-severe renal failure
* allergy to levosimendan
* lack of patient consent Pregnancy or status of lactating
* Fertile women who do not use relevant anticonception

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Juhl-Olsen, M.D., Principal Investigator — Department of Anaesthesiology
Locations (1):
- Department of Anaesthesiology, Århus N, Central Jutland, Denmark

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levosimendan | Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levosimendan | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 76 [69 to 87] | 73 [73 to 85] | 74 [69 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  Denmark | 10 | 10 | 10

OUTCOME MEASURES:

1. Primary Outcome: E/E'(Unitless)
Description: Ration between early transmitral flow (E) and mitral annular tissue velocity(E'). This ratio is an echocardiographic index of diastolic function
Time Frame: 4 hours before operation until 21 hour after operation
Measure: Median (Full Range); unit: Unitless
Arm/Group | Levosimendan | Placebo
Number analyzed (Participants) | 10 | 10
Unitless | 12.6 [8.9 to 24.6] | 13.7 [8.4 to 28.1]

2. Secondary Outcome: Isovolumetric Relaxation Time (IVRT) (s)
Description: Transthoracic measure of the time from aortic valve closure until mitral valve opening. A measure of diastolic function
Time Frame: 4 hours before surgery until 1 hour before operation
Reporting Status: Not Posted

3. Secondary Outcome: Ejection Fraction (Per Cent)
Description: Transeosophageal echocardiography: Measure of systolic function
Time Frame: At start of operation until end of operation, approximately 3 hours
Reporting Status: Not Posted

4. Secondary Outcome: Cardiac Index (l/Min/m2)
Description: Invasive measurement measuring the cardiac output divided by calculated body surface area (DuBois formula)
Time Frame: 4 hours before operation until 1 hour before operation
Reporting Status: Not Posted

5. Secondary Outcome: Central Venous Pressure (mmHg)
Description: Invasive measurement of pressure in the vena cava
Time Frame: 4 hours before operation until 1 hours before operation
Reporting Status: Not Posted

6. Secondary Outcome: Pulmonary Artery Pressures (mmHg)
Description: Invasive measurement of mean pressure in the pulmonary artery
Time Frame: 4 hours before operation until 1 hour before operation
Reporting Status: Not Posted

7. Secondary Outcome: Systemic Arterial Pressure (mmHg)
Description: Invasive measurements of arterial mean pressure
Time Frame: 4 hours before operation until 1 hour before operation
Reporting Status: Not Posted

8. Secondary Outcome: N-terminal Pro Brain Natriuretic Peptide (NT proBNP)(pg/ml)
Description: blood sample reflecting stretch of the atrium/ventricle
Time Frame: 4 hours before operation until 4 hours after operation
Reporting Status: Not Posted

9. Secondary Outcome: Troponin T (ug/l)
Description: Blood sample expressing damage to the myocytes
Time Frame: 4 hours before operation until 4 hours after operation
Reporting Status: Not Posted

10. Secondary Outcome: Lactate (mmol/l)
Description: Arterial sampling of blood lactate
Time Frame: 4 hours before operation until 4 hour after operation
Reporting Status: Not Posted

11. Secondary Outcome: Mixed Venous Oxygenation (Per Cent)
Description: Oxygen content (per cent of hemoglobin saturated) of venous blood in pulmonary artery
Time Frame: 4 hours before operation until 4 hour after operation
Reporting Status: Not Posted

12. Secondary Outcome: E/A Ratio (Unitless)
Description: TEE ratio between early (E) transmitral flow and late (A) transmitral flow. An index of diastolic function althought not validated properly yet when measured from the oesophagus
Time Frame: At the start of operation until the end of operationon, approximately 3 hours
Reporting Status: Not Posted

13. Secondary Outcome: Regional Longitudinal Strain (Unitless)
Description: Transoesophageal echocardiographic (TEE) measure of systolic function. At this time not validated properly against acknowledged indices of systolic function.
Time Frame: At the start of operation until the end of operation, approximately 3 hours
Reporting Status: Not Posted

14. Secondary Outcome: Need for Conventional Inotropical Agents
Description: Conventional inotropics are comprised of all inotropics acting primarily through alfa- or beta- stimulation.
Time Frame: From start of operation until 5 days after operation
Reporting Status: Not Posted

15. Secondary Outcome: Intravenous Fluid Requirement (l)
Description: Total volume of intravenous fluid required including blood products.
Time Frame: Within 24 hours from start of operation
Reporting Status: Not Posted

16. Secondary Outcome: Operation Time (Minutes)
Time Frame: From "knife start" until "knife end", approximately 3 hours
Reporting Status: Not Posted

17. Secondary Outcome: Time on Heart-lung Machine (Minutes)
Time Frame: From time of cardioplegia until selfsufficient cardiac action, approximately 1 hour
Reporting Status: Not Posted

18. Secondary Outcome: Intubation Time (Minutes)
Description: Total time intubated including time of operation and in the intensive care ward
Time Frame: From intubation until extubation, approximately 6 hours
Reporting Status: Not Posted

19. Secondary Outcome: Postoperative Admission Time at Intensive Care Unit (Hours)
Description: Total admission time in the intensive care after operation
Time Frame: From admission to the intensive care unit until discharge from intensive care unit, approximately 24 hours
Reporting Status: Not Posted

20. Secondary Outcome: No. of Patients With Adverse Events
Description: Development of Ventricular tachycardia
Time Frame: -4 hours until + 96 hours with respect to start of operation
Reporting Status: Not Posted

21. Secondary Outcome: No. of Patients With Adverse Event
Description: Development of atrial flutter/fibrillation
Time Frame: -4 hours until + 96 hours with respect to start of operation
Reporting Status: Not Posted

22. Secondary Outcome: No. of Patients With Adverse Event
Description: Need for norepinephrine as an antagonist to the vasodilatatory effect of levosimendan
Time Frame: 4 hours before operaton until 1 hour before operaton
Reporting Status: Not Posted

23. Secondary Outcome: No. of Patients With Adverse Event.
Description: Occurence of nausea
Time Frame: 4 hours before operation until 1 hour before operation
Reporting Status: Not Posted

24. Secondary Outcome: No. of Patients With Adverse Event
Description: Occurence of headache
Time Frame: 4 hours before operation until approximately 1 hour before operation
Reporting Status: Not Posted

25. Secondary Outcome: Regional Longitudinal Strain (Unitless)
Description: Index of systolic function derived from single transthoracic echocardiographic (TTE) projection
Time Frame: 4 hours before until 1 hour before start of operation
Reporting Status: Not Posted

26. Secondary Outcome: Ejection Fraction (Per Cent)
Description: TTE: Index of systolic function
Time Frame: 1 hour before until 21 hour after start of operation
Reporting Status: Not Posted

27. Secondary Outcome: Ejection Fraction (Per Cent)
Description: TTE: Index of systolic function
Time Frame: 21 hours after operation until 96 hours after start of operation
Reporting Status: Not Posted

28. Secondary Outcome: Ejection Fraction (Per Cent)
Description: TTE: Index of systolic function
Time Frame: 96 hours after operation until 6 months after operation
Reporting Status: Not Posted

29. Secondary Outcome: Regional Longitudinal Strain (Unitless)
Description: as for outcome 13
Time Frame: Froml the end of operation until approx 4 hours after operation
Reporting Status: Not Posted

30. Secondary Outcome: E/A Ratio (Unitless)
Description: as for outcome 12
Time Frame: At the end of operationon until approx 4 hours after operation
Reporting Status: Not Posted

31. Secondary Outcome: Left Ventricular Rotation (Degrees)
Description: TTE: Index of both systolic and diastolic function
Time Frame: 96 hour after operation until 6 months after operation
Reporting Status: Not Posted

32. Secondary Outcome: Mixed Venous Oxygenation (Per Cent)
Description: Oxygen content (per cent of hemoglobin saturated) of venous blood in pulmonary artery
Time Frame: 4 hours after operation until 21 hours after operation
Reporting Status: Not Posted

33. Secondary Outcome: Lactate (mmol/l)
Description: Arterial sampling of blood lactate
Time Frame: 4 hours after operation until 21 hours after operation
Reporting Status: Not Posted

34. Secondary Outcome: Troponin T (ug/l)
Description: Blood sample expressing damage to the myocytes
Time Frame: 4 hours after operation until 21 hours after operation
Reporting Status: Not Posted

35. Secondary Outcome: Troponin T (ug/l)
Description: Blood sample expressing damage to the myocytes
Time Frame: 21 hours after operation until 96 hours after operation
Reporting Status: Not Posted

36. Secondary Outcome: N-terminal Pro Brain Natriuretic Peptide (NT proBNP)(pg/ml)
Description: blood sample reflecting stretch of the atrium/ventricle
Time Frame: 4 hours after operation until 21 hours after operation
Reporting Status: Not Posted

37. Secondary Outcome: N-terminal Pro Brain Natriuretic Peptide (NT proBNP)(pg/ml)
Description: blood sample reflecting stretch of the atrium/ventricle
Time Frame: 21 hours after operation until 96 hours after operation
Reporting Status: Not Posted

38. Secondary Outcome: Systemic Arterial Pressure (mmHg)
Description: Invasive measurements of arterial mean pressure
Time Frame: 1 hour before operation until start of operation
Reporting Status: Not Posted

39. Secondary Outcome: Systemic Arterial Pressure (mmHg)
Description: Invasive measurements of arterial mean pressure
Time Frame: Start of operation until the end of operation, approximately 3 hours
Reporting Status: Not Posted

40. Secondary Outcome: Systemic Arterial Pressure (mmHg)
Description: Invasive measurements of arterial mean pressure
Time Frame: End of operation until approx 4 hours after operation
Reporting Status: Not Posted

41. Secondary Outcome: Systemic Arterial Pressure (mmHg)
Description: Invasive measurements of arterial mean pressure
Time Frame: 4 hours after operation until 21 hours after operation
Reporting Status: Not Posted

42. Secondary Outcome: Pulmonary Artery Pressures (mmHg)
Description: Invasive measurement of mean pressure in the pulmonary artery
Time Frame: 1 hour before operation until start of operation
Reporting Status: Not Posted

43. Secondary Outcome: Pulmonary Artery Pressures (mmHg)
Description: Invasive measurement of mean pressure in the pulmonary artery
Time Frame: Start of operation until end of operation, approximately 3 hours
Reporting Status: Not Posted

44. Secondary Outcome: Pulmonary Artery Pressures (mmHg)
Description: Invasive measurement of mean pressure in the pulmonary artery
Time Frame: End of operation until approx 4 hours after operation
Reporting Status: Not Posted

45. Secondary Outcome: Pulmonary Artery Pressures (mmHg)
Description: Invasive measurement of mean pressure in the pulmonary artery
Time Frame: 4 hours after operation until 21 hours after operation
Reporting Status: Not Posted

46. Secondary Outcome: Regional Longitudinal Strain (Unitless)
Description: Index of systolic function derived from single transthoracic echocardiographic (TTE) projection
Time Frame: 1 hour before start of operation until 21 hours after operation
Reporting Status: Not Posted

47. Secondary Outcome: Regional Longitudinal Strain (Unitless)
Description: Index of systolic function derived from single transthoracic echocardiographic (TTE) projection
Time Frame: 21 hours after operation until 96 hours after operation
Reporting Status: Not Posted

48. Secondary Outcome: Regional Longitudinal Strain (Unitless)
Description: Index of systolic function derived from single transthoracic echocardiographic (TTE) projection
Time Frame: 96 hours after operation until 6 months after operation
Reporting Status: Not Posted

49. Secondary Outcome: Central Venous Pressure (mmHg)
Description: Invasive measurement of pressure in the vena cava
Time Frame: 1 hour before operation until start of operation
Reporting Status: Not Posted

50. Secondary Outcome: Central Venous Pressure (mmHg)
Description: Invasive measurement of pressure in the vena cava
Time Frame: Start of operation until end of operation, approximately 3 hours
Reporting Status: Not Posted

51. Secondary Outcome: Central Venous Pressure (mmHg)
Description: Invasive measurement of pressure in the vena cava
Time Frame: End of operation until approx 4 hours after operation
Reporting Status: Not Posted

52. Secondary Outcome: Central Venous Pressure (mmHg)
Description: Invasive measurement of pressure in the vena cava
Time Frame: 4 hours after operation until 21 hours after operation
Reporting Status: Not Posted

53. Secondary Outcome: Peak Systolic Velocity (m/s)
Description: Tissue Doppler measure of systolic function
Time Frame: 1 hour before operation until 21 hours after operation
Reporting Status: Not Posted

54. Secondary Outcome: Peak Systolic Velocity (m/s)
Description: Tissue Doppler measure of systolic function
Time Frame: 21 hours after operation until 96 hours after operation
Reporting Status: Not Posted

55. Secondary Outcome: Peak Systolic Velocity (m/s)
Description: Tissue Doppler measure of systolic function
Time Frame: 96 hours after operation until 6 months after operation
Reporting Status: Not Posted

56. Secondary Outcome: Tricuspid Annular Plane Systolic Excursion (TAPSE) (mm)
Description: Transthoracic echocardiographic measure of systolic function
Time Frame: 1 hour before operation until 21 hours after operation
Reporting Status: Not Posted

57. Secondary Outcome: Tricuspid Annular Plane Systolic Excursion (TAPSE) (mm)
Description: Transthoracic echocardiographic measure of systolic function
Time Frame: 21 hours after operation until 96 hours after operation
Reporting Status: Not Posted

58. Secondary Outcome: Tricuspid Annular Plane Systolic Excursion (TAPSE) (mm)
Description: Transthoracic echocardiographic measure of systolic function
Time Frame: 96 hours after operation until 6 months after operation
Reporting Status: Not Posted

59. Secondary Outcome: E/A-ratio (Unitless)
Description: Transthoracic echocardiographic ratio between early (E) and late (A) transmitral blood velocities. Index of diastolic function.
Time Frame: 1 hour before operation until 21 hours after operation
Reporting Status: Not Posted

60. Secondary Outcome: E/A-ratio (Unitless)
Description: as for outcome 59
Time Frame: 21 hours after operation until 96 hours after operation
Reporting Status: Not Posted

61. Secondary Outcome: E/A-ratio (Unitless)
Description: as for outcome 59
Time Frame: 96 hours after operation until 6 months after operation
Reporting Status: Not Posted

62. Secondary Outcome: E'/A'-Ratio (Unitless)
Description: Tissue Doppler transthoracic echocardiography: Ratio between tissue velocities at the mitral plan during early (E) diastole and late (A) diastole. Index of diastolic function.
Time Frame: 1 hour before operation until 21 hours after roperation
Reporting Status: Not Posted

63. Secondary Outcome: E'/A'-Ratio (Unitless)
Description: as for outcome 62
Time Frame: 21 hours after operation until 96 hours after operation
Reporting Status: Not Posted

64. Secondary Outcome: E'/A'-Ratio (Unitless)
Description: as for outcome 62
Time Frame: 96 hours after operation until 6 months after operation
Reporting Status: Not Posted

65. Secondary Outcome: Isovolumetric Relaxation Time (IVRT) (s)
Description: Transthoracic measure of the time from aortic valve closure until mitral valve opening. A measure of diastolic function
Time Frame: 1 hour before operation until 21 hours after operation
Reporting Status: Not Posted

66. Secondary Outcome: Isovolumetric Relaxation Time (IVRT) (s)
Description: Transthoracic measure of the time from aortic valve closure until mitral valve opening. A measure of diastolic function
Time Frame: 21 hours after operation until 96 hours after operation
Reporting Status: Not Posted

67. Secondary Outcome: Isovolumetric Relaxation Time (IVRT) (s)
Description: Transthoracic measure of the time from aortic valve closure until mitral valve opening. A measure of diastolic function
Time Frame: 96 hours after operation until 6 months after operation
Reporting Status: Not Posted

68. Secondary Outcome: Ejection Fraction (Per Cent)
Description: Transeosophageal echocardiography: Measure of systolic function
Time Frame: End of operation until approx. 4 hours after operation
Reporting Status: Not Posted

69. Secondary Outcome: Isovolumetric Relaxation Time (IVRT) (s)
Description: Transeosophageal echocardiography: Time from closure of aortic valve to opening of mitral valve. Measure of diastolic function.
Time Frame: End of operation until approx. 4 hours after operation
Reporting Status: Not Posted

70. Secondary Outcome: Cardiac Index (l/Min/m2)
Description: Invasive measurement measuring the cardiac output divided by calculated body surface area (DuBois formula)
Time Frame: 1 hour before operation until start of operation
Reporting Status: Not Posted

71. Secondary Outcome: Cardiac Index (l/Min/m2)
Description: Invasive measurement measuring the cardiac output divided by calculated body surface area (DuBois formula)
Time Frame: Start of operation until end of operation, approximately 3 hours
Reporting Status: Not Posted

72. Secondary Outcome: Cardiac Index (l/Min/m2)
Description: Invasive measurement measuring the cardiac output divided by calculated body surface area (DuBois formula)
Time Frame: End of operation operation until approx. 4 hours after operation
Reporting Status: Not Posted

73. Secondary Outcome: Cardiac Index (l/Min/m2)
Description: Invasive measurement measuring the cardiac output divided by calculated body surface area (DuBois formula)
Time Frame: 4 hours after operation until 21 hours after operation
Reporting Status: Not Posted

74. Secondary Outcome: Inflammatory Parameters
Description: Blood sample values of pro- and antiinflammatory mediators
Time Frame: 4 hours before operation until 21 hours after operation
Reporting Status: Not Posted

75. Secondary Outcome: Inflammatory Parameters
Description: Blood sample values of pro- and antiinflammatory mediators
Time Frame: 21 hours after operation until 96 hours after operation
Reporting Status: Not Posted

76. Secondary Outcome: E/A-ratio (Transoesophageal)
Description: Transoesophageal echocardiographic measure of diastolic heart function
Time Frame: from start of operation until end of operation, approximately 3 hours
Reporting Status: Not Posted

77. Secondary Outcome: E/A-ratio (Transoesophageal)
Description: Transoesophageal echocardiographic measure of diastolic heart function
Time Frame: from end of operation until approximately 4 hours after operation
Reporting Status: Not Posted

78. Secondary Outcome: Urine Clearance
Description: Urine analysis. Measure of kidney function.
Time Frame: from start of operation until 24 hours after operation
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Levosimendan | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levosimendan (N=10) | Placebo (N=10)
Postoperative atrial fibrillation (Cardiac disorders) | 9 (10) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes